CLINICAL TRIAL: NCT06285370
Title: An Open-Label, Multicenter, Single Arm Study to Evaluate the Efficacy and Safety of Anti-CCR4 Monoclonal Antibody Mogamulizumab (KW-0761) in Chinese Subjects With Mycosis Fungoides or Sézary Syndrome Previously Treated With Systemic Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of KW-0761 in Chinese Subjects With Mycosis Fungoides or Sézary Syndrome Previously Treated With Systemic Therapy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-CN001; CTR20230672 (Other: National Medical Products Administration)
Record Dates: First submitted 2023-08-16; First posted 2024-02-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: mycosis fungoides/sézary syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — mogamulizumab

STUDY DESIGN:
Intervention Model Description: This is an open-label, multicenter, single arm study.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KW-0761 (Experimental): Patients will receive KW-0761 in this arm
  Interventions: Drug: Mogamulizumab

INTERVENTIONS:
Drug: Mogamulizumab — Mogamulizumab will be administered at the dose of 1.0 mg/kg as an intravenous (iv) infusion over at least 1 hour on Days 1, 8, 15, and 22 of Cycle 1 and on Days 1 and 15 of subsequent cycles. Each treatment cycle is set as 28 days. Subjects will continue the treatment of mogamulizumab until any of the criteria for study withdrawal is met.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of mogamulizumab (KW-0761) in chinese subjects with mycosis fungoides or sézary syndrome previously treated with systemic therapy

DETAILED DESCRIPTION:
This is an open-label, multicenter, single arm study. This study consists of three parts: the Pretreatment Period, the Treatment Period, and the Follow-up Period. Subjects who meet all of eligibility criteria by the screening examination will be enrolled into the study, and start treatment with mogamulizumab within 30 days after obtaining consent. Mogamulizumab will be administered at the dose of 1.0 mg/kg as an intravenous (iv) infusion over at least 1 hour on Days 1, 8, 15, and 22 of Cycle 1 and on Days 1 and 15 of subsequent cycles. Each treatment cycle is set as 28 days. Subjects will continue the treatment of mogamulizumab until any of the criteria for study withdrawal is met. After stopping treatment, the end-of treatment examination will be conducted within 30 days after the last dose.The primary efficacy analysis will be conducted once all subjects terminate treatment by the confirmation of PD/drug intolerance/unacceptable toxicity or 12 months after the date of the first mogamulizumab administration of the last subject of entire study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated ethics committee (EC) approved informed consent form in accordance with regulatory and institutional guidelines. Written informed consent must be obtained prior to performing any study-related procedure.
2. Male and female Chinese subjects ≥18 years of age at the time that written informed consent is obtained.
3. Histologically confirmed diagnosis of MF or SS;
4. Stage IB, IIA, IIB, III, and IV.
5. Patients who have failed at least one prior systemic therapy. Systemic therapy includes, for example, interferon, denileukin diftitox, retinoid, photopheresis, anti-neoplastic chemotherapy, methotrexate, and Histone deacetylase (HDAC) inhibitor.

   - Ultraviolet light therapy (Psoralen plus ultraviolet A [PUVA], ultraviolet B [UVB] etc), systemic steroid monotherapy, topical steroid or other topical agents, and any radiation are not considered to be a systemic therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1.
7. The subject has resolution of all clinically significant toxic effects of prior cancer therapy to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE, ver. 5.0) excluding the specifications required in 8, 9, and 10 below.
8. Adequate hematological function:

   * absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * platelets ≥ 100.0 × 10^9/L;
   * in subjects with known bone marrow involvement, ANC must be ≥ 1.0 × 10^9/L and platelets ≥ 75.0 × 10^9/L.
9. Adequate hepatic function:

   * Total bilirubin ≤ 1.5 times the specific institutional upper limit of normal (ULN);
   * aspartate transaminase (AST) and alanine transaminase (ALT) each ≤ 2.5 × ULN or ≤ 5.0 × ULN in the presence of known hepatic involvement by CTCL.
10. Adequate renal function:

    - serum creatinine (SCr) ≤ 1.5 × ULN, or calculated creatinine clearance (CCr)> 50 mL/min using the Cockcroft-Gault formula. To calculate CCr, the body weight and SCr results on the same day should be used.
11. Patients with MF and a known history of non-complicated staphylococcus infection/colonization are eligible provided they continue to receive stable doses of prophylactic antibiotics.
12. Women of childbearing potential must have a negative pregnancy test within 7 days prior to receiving study medication.
13. Women of childbearing potential (WOCBP)* and fertile men who consent to practice contraception using highly effective methods during a period from the day providing her consent to the end of the study (for women) or from the start of IP administration to the end of the study (for men). WOCBP shall have a negative pregnancy test result in the screening examination and a negative pregnancy test result in the pre-dose examination at Day 1.

    * WOCBP do not include women who underwent permanent contraception, postmenopausal women (in the case of the absence of menstruation for 12 months or more regardless of other medical reasons and serum follicle stimulating hormone (FSH) level >40 mIU/mL) and women who are anatomically incapable of becoming pregnant.

Exclusion Criteria:

1. Current evidence of large cell transformation (LCT). Patients with clinical features suggestive of LCT are recommended to have a biopsy performed within 4 months prior to Cycle 1 Day 1 to rule out transformed disease. Patients with a history of LCT but without current aggressive disease and no current evidence of LCT on pathology in skin or lymph nodes are eligible.
2. Diagnosed with a malignancy other than MF/SS in the past 2 years from the time that written informed consent is obtained. However, subjects with non-melanoma skin cancers, melanoma in situ, localized cancer of the prostate with current prostate-specific antigen of < 0.1 ng/mL, treated thyroid cancer or cervical carcinoma in situ, or ductal/lobular carcinoma in situ of the breast within the past 2 years may be enrolled as long as there is no current evidence of disease.
3. Clinical evidence of central nervous system metastasis.
4. Psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit compliance with study requirements.
5. Significant uncontrolled intercurrent illness including, but not limited to:

   * uncontrolled infection requiring antibiotics;
   * clinically significant cardiac disease (Class III or IV of the New York Heart Association [NYHA] classification);
   * unstable angina pectoris;
   * angioplasty, stenting, or myocardial infarction within 6 months;
   * uncontrolled hypertension (systolic blood pressure [BP] > 160 mmHg or diastolic BP>100 mmHg, found on 2 consecutive measurements separated by a 1-week period) despite 2 antihypertensive medications;
   * clinically significant cardiac arrhythmia;
   * uncontrolled diabetes.
6. Known or tests positive for human immunodeficiency virus (HIV) or history of HIV infection, or hepatitis C disease or history of hepatitis C infection.
7. Tests positive for hepatitis B virus surface (HBs) antigen or both HBc antibody and hepatitis B virus (HBV)-DNA positive (over the lower limit of quantification);

   - Patients with HBs antibody positive due to a hepatitis B vaccine will be allowed to participate in this trial.
8. Active herpes simplex or herpes zoster. Patients on prophylaxis for herpes who started taking medication at least 30 days prior to the pretreatment visit, have no signs of active infection, and whose last active infection was more than 6 months ago may enter the study, and should continue to take the prescribed medication for the duration of the study.
9. Experienced allergic reactions to monoclonal antibodies or other therapeutic proteins.
10. Known active autoimmune disease (e.g., Graves' disease; systemic lupus erythematosus; rheumatoid arthritis; Crohn's disease; psoriasis).
11. Is pregnant (confirmed by beta human chorionic gonadotrophin [β-HCG]) or lactating.
12. Prior treatment with mogamulizumab.
13. Have had any therapy directed against the subject's underlying cancer or any investigational medications within 4 weeks of registration (skin directed treatments, including topicals and radiation within 2 weeks of registration treatment).
14. Subjects on a stable dose of a low dose systemic corticosteroid (≤ 20 mg prednisone equivalent) for at least 4 weeks prior to the registration may continue use although the investigator should attempt to taper the use to the lowest dosage tolerable while on study.
15. Subjects on a stable dose of medium or low potency topical corticosteroids for at least 4 weeks prior to the registration may continue use at the same dose, although the investigator should attempt to taper the use to the lowest dosage tolerable while on study.
16. History of allogeneic transplant.
17. Autologous hematopoietic stem cell transplant within 90 days of the screening.
18. Patients on any immunomodulatory drug for concomitant or intercurrent conditions or who have received any of these agents within 4 weeks of registration, including but not limited to the following, will be excluded: low-dose or oral methotrexate, azathioprine, iv immunoglobulin, low-dose or oral cyclophosphamide, cyclosporine, mycophenolate, infliximab, etanercept, leflunomide, adalimumab, lenalidomide, abatacept, rituximab, anakinra, interferon-β, interleukin-2, and natalizumab.
19. Anyone otherwise considered unsuitable participation in the study by the investigator or subinvestigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  The ORR was defined as the count of subjects who had a confirmed CR or PR, defined as documented CR or PR per Global Composite Response Score that was confirmed by a subsequent observation at least 4 weeks later. Overall Response Rate was determined based on the response in all compartments (lymph nodes, skin, peripheral blood, and viscera), referencing Olsen, 2011 as follows: Complete Response (CR) = complete disappearance of all clinical evidence of disease; Partial Response (PR) = regression of measurable disease; Stable Disease (SD) = failure to attain CR, PR, or PD; Progressive Disease (PD) = PD in any compartment; Relapse = recurrence of disease in prior CR in any compartment.

SECONDARY OUTCOMES:
Skin disease response rate; | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  Skin disease will be evaluated using the modified SWAT. The detailed response criteria (CR, PR, PD, SD) is defined in Olsen 2011. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects
Lymth nodes response rate | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  Lymph nodes status will be evaluated by enhanced computed tomography (CT）. The detailed response criteria (CR, PR, PD, SD) is defined in Olsen 2011. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects
Visceral metastases response rate; | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  Visceral disease status will be evaluated by enhanced computed tomography (CT）. The detailed response criteria (CR, PR, PD, SD) is defined in Olsen 2011. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects.
Blood disease response rate; | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  The response in blood will be assessed by flow cytometry. The detailed response criteria (CR, PR, PD, SD) is defined in Olsen 2011. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects.
Progression Free Survival | Up to 32 months.
  PFS is defined as the time from the first day of a treatment until documented progression or death.
  Progression was defined based on Olsen (2011).
Duration of response (DOR) | Up to 32 months.
  The DOR is defined as the time from the date that criteria for CR or PR are met (whichever is first recorded) until the first date that PD or death is objectively documented. Subjects who still continue response at the time of analysis will be censored at the day of their last tumor assessment (from any compartment).
Time to response (TTR) | Up to 29 months.
  TTR is defined as the time from the date of first dose to the date that criteria for CR or PR are met (whichever is first recorded). Subjects who do not meet response criteria will be censored at the day of their last tumor assessment (from any compartment).
Response rate of lymph node evaluated by Lugano 2014. | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  Subjects will be evaluated for response in lymph node based on Lugano 2014 criteria. Disease status will be evaluated by enhanced computed tomography (CT）. The detailed response criteria (CR, PR, PD, SD) is defined in Lugano 2014. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects.
Response rate of viscera evaluated by Lugano 2014 criteria. | At the end of each cycle (each cycle is 28 days) until progression up to 29 months;
  Subjects will be evaluated for response in viscera based on Lugano 2014 criteria. Disease status will be evaluated by enhanced computed tomography (CT）. The detailed response criteria (CR, PR, PD, SD) is defined in Lugano 2014. Complete response (CR) or partial response (PR) will be regarded as response. Response rate is calculated by Subjects who confirmed response/Total subjects.

OTHER OUTCOMES:
To evaluate pharmacokinetics (plasma mogamulizumab concentration) of mogamulizumab. | Day 1 (Before infusion and at the end of the infusion), Day 8, Day 15, Day 22, Days 28 in Cycle 1; Day 15, Days 28 in Cycle 2 and 3; Days 28 in Cycle 4, 6, 8, 10, 12; Last visit. Each cycle is 28 days.
To evaluate immunogenicity (anti-mogamulizumab antibody) of mogamulizumab. | Day 1, Days 28 in Cycle 1; Days 28 in Cycle 2, 3, 4, 6, 8, 10, 12; Last visit. Each cycle is 28 days.
To evaluate the effects of skin disease on health-related Quality of Life (HRQoL) -Skindex 29. | Day 1, Days 28 in Cycle 1; Days 28 in odd cycles (Cycle 3, 5, 7, 9, 11, 13, 15…); Last visit. Each cycle is 28 days.
  Skindex-29 rates 29 items assessing 3 domains (emotions, symptoms, & functioning) on a linear scale from 0 (never) to all the time (100). Higher scores = higher impact of skin disease.
The incidence and frequency of treatment-related adverse events (TEAEs) and drug-related TEAEs as assessed by CTCAE v5.0. | Information from the date of the subject's signing the ICF until 90 days after the last dose or initiation of alternative therapy, whichever comes first will be recorded.
  An AE can be any unfavorable or unintended signs (including any abnormal laboratory findings), symptoms, or disease that occurred after subject's signing the ICF.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Chinese Academy of Medical Sciences
Locations (8):
- China (8):
  - Peking University First Hospital, Department of Dermatology and Venereology, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Department of Medical Oncology, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhengzhou University, Henan, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.
URL: https://vivli.org/ourmember/kyowa-kirin/